# Cover Letter:

Official project title:

Technological-based Personalized Care Intervention for Supporting Older People with Diabetes Mellitus

Funding source: HKMU R&D Fund

NCT number: HE-RD/2023/1.11

Document updated date: 12/09/2023

Document updated date: 12/09/2023

# **Information Sheet**

### TITLE OF THE STUDY

Technological-based Personalized Care Intervention for Supporting Older People with Diabetes Mellitus

### INTRODUCTORY SENTENCE

You are invited to participate in a research study conducted by Associate Professor, Dr. Law Pui Sze Queenie from the School of Nursing and Health Studies of Hong Kong Metropolitan University (HKMU).

### PURPOSE OF THE STUDY

This study will aim to investigate the effect of Technological-based Personalized Care Intervention for Supporting Older People with Diabetes Mellitus. The result may provide indication to health care professionals and population at risk to integrate non-invasive technology into the management of diabetes.

### **PROCEDURES**

The study would be last for eight weeks. You are invited to screen for the inclusion criteria and sign a consent form before participation in this study. You are invited to have your HbA1C level measured using a point-of-care test (POCT). Secondary outcomes will be lipid panel, blood glucose, blood pressure, body mass index, breath and blood ketone respectively and complete a set of psychometric questionnaires, which will take you about 45 minutes, before the intervention, start of the intervention (T0), and again at 8 weeks (T1) to determine their short-term effects.

The proposed study will adopt a RCT with two treatment arms to clarify the effects of non-invasive blood glucose device on blood glucose monitoring. The two arms will be the non-invasive blood glucose monitoring (arm 1) and traditional self-monitoring (arm 2) as a control. The interventions are referring to either non-invasive blood glucose monitoring or traditional self-monitoring control group. If you are assigned to non-invasive blood glucose monitoring group, you will receive non-invasive blood glucose monitoring and phone consultation and follow-up for eight weeks. If you are traditional self-monitoring control group, you are required to care as traditional self-monitoring of blood glucose and phone consultation and follow-up for eight weeks.

# POTENTIAL RISKS/STRESS/PAIN/DISCOMFORTS/OTHER FACTORS AND THEIR MINIMIZATION

The testing should not result in any undue discomfort. The possible minor pain is the finger-prink blood test.

### POTENTIAL BENEFITS

Participation in this research project is free of charge including phone counselling sessions and body measurement tests.

### PARTICIPATION AND WITHDRAWAL

Your participation is voluntary and that you can choose to withdraw from the study at any time you want without any penalty or negative consequences.

Document updated date: 12/09/2023

### **CONFIDENTIALITY**

All information related to you will remain confidential and will be identifiable by codes only known to the researchers. The information you provide as part of the project is the research data. Any research data from which you can be identified is known as personal data. Personal data does not include data where the identity has been removed (anonymous data). We will minimize our use of personal data in the study as much as possible. The researcher team will have access to personal data and research data for the purposes of the study. Responsible members of HKMU may be given access to data for monitoring and/or audit of the study to ensure that the research is complying with applicable regulations.

### **OUESTIONS AND CONCERNS**

If you have any questions or concerns about the research study, please feel free to contact Associate Professor, Dr. Queenie Law of HKMU at 3970 2974 or via email: qlaw@hkmu.edu.hk. If you have questions about your rights as a participant of this research study, please contact the Research Ethics Committee of HKMU at 27686251.

## **Consent Form**

Hong Kong Metropolitan University School of Nursing and Health Studies

Technological-based Personalized Care Intervention for Supporting Older People with Diabetes Mellitus

I have read and understand the information provided about the above study. I agree to participate in this study.

| Name of participant | Signature of participant | Date |
|----------------------|---------------------------|------|
| Name of investigator | Signature of investigator | Date |

Document updated date: 12/09/2023